CLINICAL TRIAL: NCT05719259
Title: POS-VAP: Perpetual Observational Study - Ventilator Associated Pneumonia
Brief Title: Perpetual Observational Study - Ventilator Associated Pneumonia
Acronym: POS-VAP
Status: Recruiting | Type: Observational
Sponsor: European Clinical Research Alliance for Infectious Diseases (ECRAID) (Other)
Collaborators: Centre Hospitalier Universitaire Dupuytren de Limoges (CHUL) (Unknown); Université de Genève (UNIGE) (Unknown); University Medical Center Utrecht (UMCU) (Unknown)
Responsible Party: Sponsor
Other Study IDs: ECRAID-Base POS-VAP
Record Dates: First submitted 2022-07-06; First posted 2023-02-08 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Ventilator Associated Pneumonia; Hospital Acquired Infection; Mechanical Ventilation; Intensive Care Unit
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days

GROUPS / COHORTS (3):
- Enrolled population: All patients meeting eligibility criteria (Adult patients, under a documented or expected time under mechanical ventilation of at least >48h) and providing one of:
  * Informed consent
  * Hospital level consent
  * Non-objection notice
  * Waiver of consent
- VAP population: Subset of the enrolled population fulfilling U.S. Food and Drug Administration (FDA) criteria for VAP diagnosis at any time during the follow up
- Microbiologically evaluable VAP population: Subset of the VAP population with a documented causative agent (bronchoalveolar lavage [BAL], endotracheal aspirate [ETA], blood sample, sputum, or pleural fluid) within 48 hours from VAP diagnosis

SUMMARY:
Ventilator-Associated Pneumonia (VAP) is a bacterial respiratory infection that patients in the Intensive Care Unit (ICU) often get when they cannot breathe for themselves and require mechanical ventilation. It is linked to higher chances of death, a longer stay in the hospital, higher costs, and the use of more antibiotics.

Options to help prevent or treat this disease are in development and will require evaluation in future clinical trials.

The goal of POS-VAP is to build and continuously train a network of ICUs to be prepared for doing these trials, to facilitate their execution.

DETAILED DESCRIPTION:
Ventilator associated pneumonia (VAP) is one of the most frequent healthcare associated infections in the Intensive Care Unit (ICU) and a significant burden among ICU patients under invasive mechanical ventilation (IMV).

Several preventive and therapeutic treatment options are being developed in the field of VAP that will require evaluation in future randomized controlled trials (RCTs).

RCTs are the gold standard for evaluating medical interventions but are difficult to perform in a population at risk of, or with, VAP.

These trials are challenging since it is difficult to recruit a large enough volume of high-quality centers to achieve the required number of recruited patients, especially if the focus is on specific patient groups (e.g., VAP due to a specific pathogen), for which site selection can be even more challenging and time consuming. There is a need for a well-organized and well-trained international network of ICUs focusing on VAP research that enables efficient execution of RCTs on diagnostic, preventive and curative interventions in this population.

Through a Perpetual Observational Study (POS) we can provide quick access to a network of sites that fulfill pre-specified criteria. Additionally, the structured network of POS sites within ECRAID will maintain continuous activity to carry out observational studies in this specific field, implementing informed consent (where required), increasing quality and efficiency, and facilitating contracting.

ELIGIBILITY:
Inclusion criteria:

* Age≥18 years
* At risk of acquiring VAP during ICU stay, defined as:
* Requiring admission or being admitted to the ICU.
* Expected or documented to be under IMV for more than 48 hours.
* Consent, either a written informed consent given by the study patient in full medical, psychological, cognitive, social or legal capacity to give an informed consent, or, if not possible, by a Legally Authorized Representative of the study patient OR any applicable locally accepted form of consent OR consent waiver allowing data collection and sharing of data according to ECRAID's principles

Exclusion Criteria:

* Death is deemed to be imminent or inevitable during this hospital admission AND one or more of the patient, substitute decision maker or attending physician are not committed to full active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to an ICU, who are under IMV and documented or expected to be under IMV for more than 48 hours are eligible to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of research sites recruiting patients | 4 years
  POS-VAP' overarching objective is to build a sustainable European clinical research network of ICUs that serves as platform to facilitate observational and randomized VAP research activities.
  This objective will be measured by in three ways:
  1. Total number of sites in the POS-VAP network that actively recruit patients
Number of patients recruited in the study | 4 years
  2. Total number of patients in the POS-VAP network per analysis population (enrolled population, VAP population and microbiologically evaluable VAP population).
Number of studies implemented through the network | 4 years
  3. Total number of implemented observational studies and RCTs (stratified by domain: prevention, diagnosis and treatment).

SECONDARY OUTCOMES:
Proportion of sites recruiting for an study implemented through the network | 4 years
  Average proportion of sites actively recruiting for at least one embedded study at any time during the study period, overall and stratified by observational and interventional embedded studies.
Proportion of patients enrolled through POS-VAP that are part of a preventive study implemented through the network | 4 years
  Proportion (%) of POS-VAP enrolled population included in an embedded preventive study, stratified by observational and interventional embedded studies.
Proportion of patients enrolled through POS-VAP that are part of a diagnostic study implemented through the network | 4 years
  Proportion (%) of POS-VAP enrolled population included in an embedded diagnostic study, stratified by observational and interventional embedded studies.
Proportion of VAP patients enrolled through POS-VAP that are part of a treatment study implemented through the network | 4 years
  Proportion (%) of POS-VAP VAP population enrolled in at least one embedded treatment study with clinical outcome after VAP as endpoint, stratified by observational and interventional embedded studies.

OTHER OUTCOMES:
Incidence of VAP per 1000 ventilation days | 4 years
  Incidence of VAP per 1000 ventilation days, measured among the Enrolled population, overal and per site
ICU mortality rate in non-VAP patients | 4 years
  ICU mortality, measured among the Enrolled population not developping VAP, overal and per site
Time from intubation until VAP diagnosis (days) | 4 years
  Time from start of invasive mechanical ventilation (IMV) until VAP diagnosis (days), measured among the VAP population, overall and per site
Time under IMV after VAP diagnosis (days) | 4 years
  Time under IMV after VAP diagnosis (days), measured among the VAP population, measured overall and per site
IMV-free days from VAP diagnosis till day 28 after VAP diagnosis (days) | 4 years
  IMV-free days from VAP diagnosis till day 28 after VAP diagnosis (days), measured among the VAP population, overall and per site
Length of ICU stay after VAP diagnosis (days) | 4 years
  Length of ICU stay after VAP diagnosis (days), measured among the VAP population, overall and per site
All-cause mortality at day 28 after VAP diagnosis (%) | 4 years
  All-cause mortality at day 28 after VAP diagnosis (%), measured among the VAP population, overall and per site
ICU mortality rate | 4 years
  Mortality rate at ICU discharge, measured among the VAP population, overall and per site
Resolution of signs and symptoms of VAP between days 7 and 10 from VAP diagnosis (%) | 4 years
  Resolution of signs and symptoms of VAP between days 7 and 10 from VAP diagnosis (%), measured among the VAP population, overall and per site

CONTACTS AND LOCATIONS:
Locations (35):
- University Hospital of Trauma, Tirana, Albania
- Belgium (5):
  - Cliniques Universitaires Saint-Luc UCL, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Hôpital de Jolimont, La Louvière
  - Centre Hospitalier Universitaire de Liège, Liège
  - Clinique Saint Pierre Ottignies, Ottignies-Louvain-la-Neuve
- Croatia (3):
  - Clinical Hospital Center Rijeka, Rijeka
  - General Hospital "Dr. Josip Benčević" Slavonski Brod, Slavonski Brod
  - University Hospital for Infectious Diseases, Zagreb
- Czechia (2):
  - University Hospital Kralovske Vinohrady, Brno-Vinohrady
  - University Hospital Motol, Prague
- France (6):
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre Hospitalier Universitaire Dijon Bourgogne, Dijon
  - Centre Hospitalier de Le Mans, Le Mans
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire Dupuytren of Limoges, Limoges
  - Centre Hospitalier Universitaire de Tours, Tours
- University Hospital Leipzig, Leipzig, Germany
- Greece (4):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Evangelismos General Hospital of Athens, Athens
  - Sotiria Thoracic Diseases Hospital of Athens, Athens
  - General University Hospital of Larissa, Larissa
- IRCCS Ospedale Policlinico Gemelli, Roma, Italy
- Netherlands (2):
  - Deventer Ziekenhuis, Deventer
  - University Medical Center Utrecht, Utrecht
- Romania (2):
  - Central Military Emergency University Hospital Dr. Carol Davila, Bucharest
  - Elias University Emergency Hospital, Bucharest
- University Clinical Center of Serbia, Belgrade, Serbia
- Spain (4):
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - IMED Valencia, Burjassot, Valencia
  - Vall d'Hebrón University Hospital, Barcelona
- United Kingdom (3):
  - John V Farman Intensive Care Unit, Cambridge
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Victoria Infirmary, Newcastle

IPD SHARING:
Plan to Share IPD: Undecided
Data from this study will be used to inform future observational studies and RCTs about expected frequencies of exposures and clinical outcomes and expected recruitment rates for specific patient populations. Furthermore, the data will be used to support simulations to gain insight in the optimal design and required sample size of future RCTs as required for future embedded studies, which will be described in the appendices.

REFERENCES:
- [Background] Hassoun-Kheir N, van Werkhoven CH, Dunning J, Jaenisch T, van Beek J, Bielicki J, Butler CC, Francois B, Harbarth S, Hernandez Padilla AC, Horby P, Koopmans M, Lee J, Rodriguez-Bano J, Tacconelli E, Themistocleous Y, van der Velden AW, Bonten M, Goossens H, de Kraker MEA; ECRAID-Base consortium. Perpetual observational studies: new strategies to support efficient implementation of observational studies and randomized trials in infectious diseases. Clin Microbiol Infect. 2022 Dec;28(12):1528-1532. doi: 10.1016/j.cmi.2022.07.024. Epub 2022 Aug 5. No abstract available. PMID 35940566
- See also: Related Info — https://www.ecraid.eu/study/pos-vap